CLINICAL TRIAL: NCT05293171
Title: A Single-Dose, Randomized, Double-Blind, Placebo-Controlled, Positive-Controlled, Four-Way Crossover Study to Investigate the Effect of BL-8040 (Motixafortide) on the QTc Interval in Healthy Subjects
Brief Title: Study to Investigate the Effect of BL-8040 (Motixafortide) on the QTc Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: BL-8040.TQT.103
Record Dates: First submitted 2022-02-02; First posted 2022-03-24 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — 4-fluorobenzoyl-TN-14003; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind (in respect to BL-8040 and BL-8040-matching placebo dosing), placebo- and positive-controlled, 4-period, 4-way crossover study. On Day 1 of Period 1, subjects will be randomized to 1 of 12 treatment sequences.
  Each treatment sequence comprises 4 treatment periods. Each subject will be assigned a unique identification number upon screening. Subjects who complete the study screening assessments and meet all the eligibility criteria will be assigned a unique randomization identification number at the time of the first dosing, different from the screening number, and will receive the corresponding study drug, according to a randomization scheme.
  Subjects will receive each of the 4 Treatments in a pre-defined order according to the sequence scheme determined at randomization.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1.25 mg/kg BL-8040 + BL-8040-matching placebo administered via SC injection (Therapeutic) (Experimental): 1.25 mg/kg BL-8040 + BL-8040-matching placebo administered via SC injection (Therapeutic)
  Interventions: Drug: 1.25 mg/kg BL-8040 + BL-8040-matching placebo
- 2 mg/kg BL-8040 administered via SC injection (Supratherapeutic) (Experimental): 2 mg/kg BL-8040 administered via SC injection (Supratherapeutic)
  Interventions: Drug: 2 mg/kg BL-8040
- BL-8040-matching placebo administered via SC injection (Placebo Comparator): BL-8040-matching placebo administered via SC injection
  Interventions: Drug: BL-8040-matching placebo
- 400 mg moxifloxacin (1 x 400 mg tablet) administered orally (Active Comparator): 400 mg moxifloxacin (1 x 400 mg tablet) administered orally
  Interventions: Drug: 400 mg Moxifloxacin (1x400 mg tablet)

INTERVENTIONS:
Drug: 1.25 mg/kg BL-8040 + BL-8040-matching placebo — Administered via subcutaneous (SC) injection
  Arms: 1.25 mg/kg BL-8040 + BL-8040-matching placebo administered via SC injection (Therapeutic)
Drug: 2 mg/kg BL-8040 — Administered via subcutaneous (SC) injection
  Arms: 2 mg/kg BL-8040 administered via SC injection (Supratherapeutic)
Drug: BL-8040-matching placebo — Administered subcutaneous (SC) injection
  Arms: BL-8040-matching placebo administered via SC injection
Drug: 400 mg Moxifloxacin (1x400 mg tablet) — Administered orally
  Arms: 400 mg moxifloxacin (1 x 400 mg tablet) administered orally

SUMMARY:
The study will assess the corrected QT (QTc) effects (electrocardiogram [ECG]) of motixafortide (BL-8040) 1.25 mg/kg (therapeutic dose) and 2 mg/kg (supratherapeutic dose) following a single subcutaneous (SC) injection relative to placebo in approximately 40 healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind (in respect to BL-8040 and BL-8040-matching placebo dosing), placebo- and positive-controlled, 4-period, 4-way crossover study in healthy subjects.

A continuous 12-lead cardiodynamic ECG recording will be collected for approximately 24 hours on Day -1 of Period 1 for use in the optimized individual corrected QTc (QTcI) baseline calculations.

On Day 1 of Period 1, subjects will be randomized to 1 of 12 treatment sequences. Each treatment sequence comprises 4 treatment periods.

On Day 1 of each period, subjects will receive single-dose SC injection of BL-8040 (therapeutic or supratherapeutic dose), single-dose SC injection of BL-8040-matching placebo, or a single oral dose of moxifloxacin. Cardiodynamic readings, plasma pharmacokinetic (PK) samples, and blood pharmacodynamic (PD) samples will be collected at different time points prior to dosing and up to 24 hours postdose in each period, as appropriate.

There will be a washout period of 5-7 days between dosing in each period.

All subjects who received at least one dose of any study drug (including subjects who terminate the study early) will return to the clinical research unit (CRU) 7 ± 2 days after the last dose for follow-up procedures, and to determine if any adverse event (AE) has occurred since the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, males and females between the ages of 18 and 55 years, inclusive, at Screening.
* Body weight between 50-109 kg (inclusive) and body mass index (BMI) within 18.0-29.99 kg/m2 (inclusive) at Screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
* Current non-smokers who have not used any nicotine-containing products (chewed or smoked) or replacement products including electronic cigarettes for at least 3 months prior to first dosing.
* Women must meet one of the following criteria: a) postmenopausal; b) surgically sterile; c) of childbearing potential and practicing contraception, as described below:

  * Postmenopausal (postmenopausal women must have no menstrual bleeding for at least 1 year prior to first dosing and menopause is confirmed by follicle-stimulating (FSH) levels consistent with postmenopausal status), or
  * Surgically sterile (e.g., hysterectomy, bilateral oophorectomy, hysteroscopic sterilization) for at least 6 months prior to first dosing, or
  * Women of childbearing potential must be non-lactating and agree to either using a highly effective acceptable form of birth control (e.g., non-hormonal intrauterine device plus condom and spermicide).
* A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non-vasectomized male.)
* If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
* Understands the study procedures in the informed consent form (ICF), and is willing and able to comply with the protocol.

Exclusion Criteria:

* Past or present diseases, which, as judged by the PI or designee, may affect the outcome of this study or pose an additional risk to the subject by their participation in the study, including, but not limited to, significant medical abnormality including: psychiatric, neurologic, pulmonary, cardiac, gastrointestinal, genitourinary, renal, metabolic, endocrinologic, or autoimmune disorder.
* Is mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
* Positive result for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody at Screening.
* Family history of QTc prolongation or of unexplainable sudden death at <50 years of age.
* History or presence of any of the following:

  * sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged Fridericia corrected QT (QTcF) interval, or conduction abnormalities;
  * ischemic heart disease, symptomatic arrhythmias, or poorly controlled hypertension.
* Knowledge of any kind of cardiovascular disorder/condition known to increase the possibility of QT prolongation or history of additional risk factors for torsade de pointes (e.g., heart failure, clinically significant hypokalemia, family history of Long QT Syndrome or Brugada Syndrome) or cardiac conduction disorders.
* Any condition that may interfere with the absorption, metabolism, or elimination of the study drug.
* History of, or active, alcohol or illicit drug abuse as defined by the Diagnostic and Statistical Manual of Mental Disorders, fourth edition, manual, within 2 years prior to the first dosing. Alcohol abuse is defined as an average intake of two or more drinks (12 oz beer, 1.5 oz of hard liquor, or equivalent) per day.
* Laboratory safety test results that are outside of the normal reference ranges (unless clinically acceptable to the PI or designee) at Screening.
* Resting supine heart rate (HR) <50 bpm or >100 bpm at Screening or check-in (Day -2). Minor deviations will be acceptable if considered to be of no clinical significance by the PI or designee.
* Resting supine systolic blood pressure <90 mmHg or >140 mmHg; resting supine diastolic blood pressure <50 mmHg or >90 mmHg at Screening or check-in.
* Significant history or presence of ECG findings at Screening or check-in (Day -2), including:

  * QTcF >450 msec
  * QRS >110 msec, if >110 msec, result will be confirmed by a manual over read
  * PR >200 msec
  * Second or third-degree atrioventricular (AV) block.
* Significant history or presence of ECG findings as judged by the PI or designee at

Screening or check-in (Day -2), including:

* ECG abnormalities which interfere with accurate QT measurement
* T wave flattening or other abnormalities which in the opinion of the PI (or designee) may interfere with the analysis of QT intervals
* Any rhythm other than sinus rhythm, which is interpreted by the PI (or designee) to be clinically significant.
* Significant safety laboratory abnormalities that would place the subject at undue risk in the PI or designee's opinion, including but not limited to serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) >1.2 x upper limit of normal at Screening or check-in.
* Positive urine cotinine at Screening.
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days or 5 half-lives (whichever is longer) prior to the first dosing or likelihood that such treatment will be needed at any time during the study (unless approved in advance by the Sponsor). Medications listed in Section 11.4.2 will be allowed.
* Participation in another clinical study within 30 days prior to the first dosing. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.
* Donation of blood or blood loss >500 mL within the 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.
* Any condition or situation that, in the opinion of the PI or designee, would prevent proper evaluation of the safety, PK, and/or PD of the study drug according to the study protocol (e.g., poorly compliant subject, poor venous access, allergies to medical plastics/latex/adhesive dressing/medical tape).
* History of hypersensitivity or allergy to moxifloxacin or any study medication.
* History of tendonitis or tendon rupture with moxifloxacin or any other quinolone type drug.
* History of unexplained loss of consciousness, unexplained syncope, near drowning with hospital admission.
* Use of any marijuana product within 6 months prior to the first dosing.
* Use of illicit drugs or tetrahydrocannabinol-containing medicines within 6 months prior to the first dosing.
* Female subjects with a positive pregnancy test at Screening or check-in or lactating.
* Positive urine drug or alcohol results at Screening or check-in.
* Has tattoo(s) or scarring at or near the site of injection or any other condition which may interfere with injection site examination, in the opinion of the PI or designee.
* Subjects intending to lose weight during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Phoenix, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 healthy, adult male and female subjects were enrolled in study. The subjects were randomly assigned to 8 different treatment sequences comprising motixafortide (BL-8040) 1.25 mg/kg, motixafortide 2 mg/kg, placebo for motixafortide and moxifloxacin 400 mg in a crossover design. 3 subjects early discontinued the study and did not receive all four treatments, 35 subjects completed the study per protocol and received all four treatments.
Groups:
- ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin: 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 2 mg/kg motixafortide administered via SC injection (B) >> motixafortide-matching placebo administered via SC injection (C) >> 400 mg moxifloxacin administered orally (D)
- BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo: 2 mg/kg motixafortide administered via SC injection (B) >> 400 mg moxifloxacin administered orally (D) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> motixafortide-matching placebo administered via SC injection (C)
- CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide: Motixafortide-matching placebo administered via SC injection (C) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 400 mg moxifloxacin administered orally (D) >> 2 mg/kg motixafortide administered via SC injection (B)
- DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide: 400 mg moxifloxacin administered orally (D) >> motixafortide-matching placebo administered via SC injection (C) >> 2 mg/kg motixafortide administered via SC injection (B), 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A)
- BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin: 2 mg/kg motixafortide administered via SC injection (B) >> motixafortide-matching placebo administered via SC injection (C) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 400 mg moxifloxacin administered orally (D)
- CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide: Motixafortide-matching placebo administered via SC injection (C) >> 400 mg moxifloxacin administered orally (D) >> 2 mg/kg motixafortide administered via SC injection (B) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A)
- ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo: 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 2 mg/kg motixafortide administered via SC injection (B) >> 400 mg moxifloxacin administered orally (D) >> motixafortide-matching placebo administered via SC injection (C)
- DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide: 400 mg moxifloxacin administered orally (D) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> motixafortide-matching placebo administered via SC injection (C) >> 2 mg/kg motixafortide administered via SC injection (B)
- CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin: Motixafortide-matching placebo administered via SC injection (C) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 2 mg/kg motixafortide administered via SC injection (B) >> 400 mg moxifloxacin administered orally (D)
- ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide: 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> 400 mg moxifloxacin administered orally (D) >> motixafortide-matching placebo administered via SC injection (C) >> 2 mg/kg motixafortide administered via SC injection (B)
- BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide: 2 mg/kg motixafortide administered via SC injection (B) >> motixafortide-matching placebo administered via SC injection (C) >> 400 mg moxifloxacin administered orally (D) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A)
- DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo: 400 mg moxifloxacin administered orally (D) >> 2 mg/kg motixafortide administered via SC injection (B) >> 1.25 mg/kg motixafortide + motixafortide-matching placebo administered via SC injection (A) >> motixafortide-matching placebo administered via SC injection (C)
Period: Period 1 - First Dosing
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 5 to 7 Days
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - Second Dosing
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 5 to 7 Days
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - Third Dosing
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 5 to 7 Days
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 2 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - Forth Dosing
Arm/Group | ABCD: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Placebo, Moxifloxacin | BDAC: 2 mg/kg Motixafortide, Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo | CADB: Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin, 2 mg/kg Motixafortide | DCBA: Moxifloxacin, Placebo, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | BCAD: 2 mg/kg Motixafortide, Placebo, 1.25 mg/kg Motixafortide, Moxifloxacin | CDBA: Placebo, Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide | ABDC: 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin, Placebo | DACB: Moxifloxacin, 1.25 mg/kg Motixafortide, Placebo, 2 mg/kg Motixafortide | CABD: Placebo, 1.25 mg/kg Motixafortide, 2 mg/kg Motixafortide, Moxifloxacin | ADCB: 1.25 mg/kg Motixafortide, Moxifloxacin, Placebo, 2 mg/kg Motixafortide | BCDA: 2 mg/kg Motixafortide, Placebo, Moxifloxacin, 1.25 mg/kg Motixafortide | DBAC: Moxifloxacin, 2 mg/kg Motixafortide, 1.25 mg/kg Motixafortide, Placebo
Started | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 3 | 4
Completed | 2 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All subjects who have received at least one of the four treatments (motixafortide 1.25 mg/kg, motixafortide 2 mg/kg, placebo for motixafortide and moxifloxacin)
Arm/Group | All Subjects
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: QTc Effect of Single Subcutaneous (SC) Injections of Motixafortide (BL-8040) 1.25 mg/kg and 2 mg/kg
Description: Assessment of the QTc effects of motixafortide 1.25 mg/kg and 2 mg/kg following a single SC injection relative to placebo in healthy subjects by evaluation of the relationship between the plasma concentration of motixafortide and ΔΔQTcI (change from baseline in QTcI)
Time Frame: Cardiodynamic ECG recordings on Day 1 (day of dosing) at different time points prior to dosing and up to 24 hours post-dose in each period (each period is 24 hours long, a total of 4 periods)
Population: The analysis population is QT/QTc Population
Measure: Mean (90% Confidence Interval); unit: ms
Groups:
- 1.25 mg/kg Motixafortide (Therapeutic): 1.25 mg/kg motixafortide administered via SC injection (Therapeutic)
- 2 mg/kg Motixafortide (Supratherapeutic): 2 mg/kg motixafortide administered via SC injection (Supratherapeutic)
- Placebo: Placebo for motixafortide
- Moxifloxacin: Moxifloxacin 400 mg administered Orally
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic) | Placebo | Moxifloxacin
Number analyzed (Participants) | 34 | 36 | 34 | 36
ms
  0.25 hr Post-dose: number analyzed (Participants) | 34 | 36 | 33 | 36
  0.25 hr Post-dose | -0.6 [-2.29 to 1.04] | 1.1 [-1.60 to 3.78] | -3.0 [-4.02 to -1.95] | -1.1 [-2.34 to 0.23]
  0.5 hr Post-dose: number analyzed (Participants) | 33 | 35 | 34 | 36
  0.5 hr Post-dose | 4.0 [1.92 to 6.00] | 7.8 [4.98 to 10.68] | -1.4 [-2.31 to -0.49] | 2.7 [0.65 to 4.74]
  0.75 hr Post-dose: number analyzed (Participants) | 32 | 33 | 34 | 36
  0.75 hr Post-dose | 7.6 [4.54 to 10.69] | 11.8 [8.32 to 15.20] | -0.1 [-1.23 to 1.06] | 8.5 [6.20 to 10.78]
  1 hr Post-dose: number analyzed (Participants) | 30 | 33 | 34 | 35
  1 hr Post-dose | 8.1 [4.53 to 11.72] | 11.2 [8.02 to 14.41] | 1.2 [0.12 to 2.33] | 10.4 [8.26 to 12.57]
  1.5 hrs Post-dose: number analyzed (Participants) | 32 | 33 | 34 | 36
  1.5 hrs Post-dose | 5.3 [2.64 to 7.89] | 2.9 [0.27 to 5.48] | 1.8 [0.17 to 3.36] | 11.8 [9.71 to 13.82]
  2 hrs Post-done: number analyzed (Participants) | 28 | 31 | 30 | 32
  2 hrs Post-done | 2.4 [0.17 to 4.55] | 0.2 [-2.76 to 3.24] | 1.5 [0.00 to 2.95] | 14.7 [12.77 to 16.59]
  3 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 33 | 35
  3 hrs Post-dose | 0.3 [-1.51 to 2.20] | -1.9 [-4.15 to 0.44] | 2.4 [0.49 to 4.33] | 13.5 [11.44 to 15.47]
  4 hrs Post-dose: number analyzed (Participants) | 31 | 35 | 34 | 35
  4 hrs Post-dose | 3.3 [1.67 to 4.85] | 2.3 [-0.28 to 4.79] | 3.8 [2.16 to 5.50] | 15.0 [13.28 to 16.73]
  6 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 34 | 35
  6 hrs Post-dose | -7.2 [-10.12 to -4.28] | -9.0 [-11.08 to -6.97] | -5.5 [-7.78 to -3.15] | 2.5 [0.32 to 4.65]
  8 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 34 | 35
  8 hrs Post-dose | -3.8 [-6.52 to -1.15] | -6.5 [-8.42 to -4.49] | -3.5 [-5.39 to -1.68] | 5.7 [3.65 to 7.75]
  12 hrs Post-dose: number analyzed (Participants) | 31 | 31 | 32 | 34
  12 hrs Post-dose | -1.1 [-3.70 to 1.49] | -2.7 [-5.37 to 0.00] | 0.5 [-1.44 to 2.40] | 4.7 [2.71 to 6.67]
  16 hrs Post-dose: number analyzed (Participants) | 32 | 33 | 32 | 35
  16 hrs Post-dose | 4.3 [1.28 to 7.27] | 3.5 [0.64 to 6.37] | 5.6 [3.36 to 7.80] | 11.6 [9.88 to 13.39]
  24 hrs Post-dose: number analyzed (Participants) | 32 | 34 | 33 | 33
  24 hrs Post-dose | 0.2 [-1.88 to 2.28] | 0.1 [-1.68 to 1.88] | 1.8 [-0.07 to 3.66] | 3.7 [2.13 to 5.24]

2. Secondary Outcome: Evaluation of AEs, 12-lead Safety ECGs, Vital Signs, Clinical Laboratory Tests, and Physical Examinations.
Description: Evaluation of safety (by assessing adverse events (AEs), ECGs, vital signs, clinical lab tests, physical examination) and tolerability (by assessing AEs) of single therapeutic and supratherapeutic SC injections of motixafortide in healthy subjects as well as of placebo and moxifloxacin.
Time Frame: During the entire study. For each participant starting from Screening until End of Study Visit - approximately 1 month.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All Subjects enrolled, randomized and to the study and received at least one dose of any of the study treatments.
- 1.25 mg/kg Motixafortide: Treatment 1.25 mg/kg motixafortide administered SC 36 subjects out of the 38 enrolled in the study received motixafortide (BL-8040) 1.25mg/kg
- 2 mg/kg Motixafortide: Treatment 2 mg/kg motixafortide administered SC 37 subjects out of the 38 enrolled in the study received motixafortide (BL-8040) 2mg/kg
- Placebo SC: Placebo administered SC 36 subjects out of the 38 enrolled in the study received placebo for motixafortide (BL-8040)
- 400 mg Moxifloxacin: Treatment 400 mg moxifloxacin administered orally 36 subjects out of the 38 enrolled in the study received moxifloxacine 400mg
Arm/Group | All Subjects | 1.25 mg/kg Motixafortide | 2 mg/kg Motixafortide | Placebo SC | 400 mg Moxifloxacin
Number analyzed (Participants) | 38 | 36 | 37 | 36 | 36
Participants
  All-Cause Mortality | 0 | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0
  Non-serious Adverse Events | 38 | 36 | 37 | 22 | 12
  Safety ECG (clinically significant changes) | 0 | 0 | 0 | 0 | 0
  Vital Signs (clinically significant changes) | 3 | 1 | 0 | 2 | 0
  Clinical Laboratory Tests (clinically significant changes) | 38 | 36 | 36 | 0 | 1
  Physical Examination (clinically significant changes) | 38 | 35 | 37 | 22 | 11

3. Secondary Outcome: PK (AUC0-t and AUC0-inf) of Single Therapeutic and Supratherapeutic SC Injections of Motixafortide (BL-8040) in Healthy Subjects.
Description: Evaluation of pharmacokinetics (PK) (AUC0-t and AUC0-inf) of single therapeutic and supratherapeutic SC injections of motixafortide in healthy subjects.
Time Frame: Blood for motixafortide PK is collected prior to dosing and at 13 different timepoints following dosing up to 24 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic)
Number analyzed (Participants) | 35 | 37
ng*h/mL
  AUC0-t | 3678 (1052.0) | 6544 (2543.1)
  AUC0-inf: number analyzed (Participants) | 35 | 36
  AUC0-inf | 3738 (1056.3) | 6329 (1858.1)

4. Secondary Outcome: PK (AUC%Extrap) of Single Therapeutic and Supratherapeutic SC Injections of Motixafortide (BL-8040) in Healthy Subjects.
Description: Evaluation of PK (AUC%extrap) of single therapeutic and supratherapeutic SC injections of motixafortide in healthy subjects.
  AUC%extrap = (1 - AUC0-t/AUC0-inf) x 100
Time Frame: Blood for motixafortide PK is collected prior to dosing and at 13 different timepoints following dosing up to 24 hours
Population: PK population
Measure: Mean (Standard Deviation); unit: % AUC0-inf
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic)
Number analyzed (Participants) | 35 | 36
% AUC0-inf | 1.717 (0.70009) | 1.302 (0.59016)

5. Secondary Outcome: PK (Cmax) of Single Therapeutic and Supratherapeutic SC Injections of Motixafortide (BL-8040) in Healthy Subjects.
Description: Evaluation of PK (Cmax) of single therapeutic and supratherapeutic SC injections of motixafortide in healthy subjects.
Time Frame: Blood for motixafortide PK is collected prior to dosing and at 13 different timepoints following dosing up to 24 hours
Population: PK Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic)
Number analyzed (Participants) | 35 | 37
ng/mL | 2245 (791.11) | 3198 (1192.4)

6. Secondary Outcome: PK (Tmax) of Single Therapeutic and Supratherapeutic SC Injections of Motixafortide (BL-8040) in Healthy Subjects.
Description: Evaluation of PK (Tmax) of single therapeutic and supratherapeutic SC injections of motixafortide in healthy subjects.
Time Frame: Blood for motixafortide PK is collected prior to dosing and at 13 different time points following dosing up to 24 hours
Population: PK Population
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic)
Number analyzed (Participants) | 35 | 37
hr | 0.754 (0.1754) | 0.690 (0.2239)

7. Secondary Outcome: Effect of Single Therapeutic and Supratherapeutic SC Injections of Motixafortide (BL-8040) on Heart Rate
Description: Assessment of the effect of single therapeutic and supratherapeutic SC injections of motixafortide on Heart Rate (a non-QT interval ECG parameter) by change from baseline (in bpm).
  "Change from Baseline" at the Baseline timepoint (predosing) is defined as zero.
  Baseline was the average of the derived ECG intervals from the 3 ECG timepoints prior to dosing (-0.75, -0.5, and -0.25 hours) on Day 1.
  Descriptive statistics of ECG parameters (HR) by-timepoint analysis of Change-from-Baseline values was done.
Time Frame: ECG recording from prior to dosing (3 timepoints) until 24 hours following administration (13 timepoints after dosing)
Population: QT/QTc Population
Measure: Mean (90% Confidence Interval); unit: bpm
Arm/Group | 1.25 mg/kg Motixafortide (Therapeutic) | 2 mg/kg Motixafortide (Supratherapeutic) | Placebo | Moxifloxacin
Number analyzed (Participants) | 34 | 36 | 34 | 36
bpm
  0.25 hr Post-dose: number analyzed (Participants) | 34 | 36 | 33 | 36
  0.25 hr Post-dose | 3.1 [1.90 to 4.31] | 7.7 [5.05 to 10.38] | -0.8 [-1.79 to 0.14] | -0.7 [-1.44 to 0.11]
  0.5 hr Post-dose: number analyzed (Participants) | 33 | 35 | 34 | 36
  0.5 hr Post-dose | 9.3 [7.20 to 11.37] | 15.5 [12.63 to 18.47] | -1.0 [-2.02 to 0.00] | 0.1 [-1.01 to 1.16]
  0.75 hr Post-dose: number analyzed (Participants) | 32 | 33 | 34 | 36
  0.75 hr Post-dose | 10.6 [7.54 to 13.70] | 12.8 [9.88 to 15.73] | -2.2 [-3.28 to -1.05] | 0.8 [-0.55 to 2.12]
  1 hr Post-dose: number analyzed (Participants) | 30 | 33 | 34 | 35
  1 hr Post-dose | 6.3 [3.44 to 9.23] | 7.2 [4.57 to 9.88] | -2.8 [-3.99 to -1.66] | 0.9 [-0.48 to 2.30]
  1.5 hrs Post-dose: number analyzed (Participants) | 32 | 33 | 34 | 36
  1.5 hrs Post-dose | -1.5 [-3.49 to 0.56] | 0.9 [-1.43 to 3.26] | -4.1 [-5.42 to -2.75] | -1.9 [-2.86 to -0.87]
  2 hrs Post-dose: number analyzed (Participants) | 28 | 31 | 30 | 32
  2 hrs Post-dose | -1.6 [-3.58 to 0.39] | 1.0 [-0.74 to 2.77] | -5.9 [-7.40 to -4.37] | -1.2 [-2.31 to -0.15]
  3 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 33 | 35
  3 hrs Post-dose | -1.1 [-3.03 to 0.88] | 2.7 [0.74 to 4.69] | -5.5 [-6.90 to -4.00] | -2.6 [-3.74 to -1.52]
  4 hrs Post-dose: number analyzed (Participants) | 31 | 35 | 34 | 35
  4 hrs Post-dose | 1.1 [-1.09 to 3.27] | 5.7 [3.74 to 7.71] | -4.6 [-6.10 to -3.13] | -1.3 [-2.60 to -0.09]
  6 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 34 | 35
  6 hrs Post-dose | 9.8 [6.86 to 12.81] | 15.6 [13.14 to 17.99] | 2.0 [0.30 to 3.73] | 5.3 [3.65 to 7.02]
  8 hrs Post-dose: number analyzed (Participants) | 32 | 35 | 34 | 35
  8 hrs Post-dose | 5.9 [2.80 to 9.09] | 11.4 [8.93 to 13.88] | -1.6 [-3.35 to 0.17] | 2.4 [0.92 to 3.91]
  12 hrs Post-dose: number analyzed (Participants) | 31 | 31 | 32 | 34
  12 hrs Post-dose | 10.8 [8.21 to 13.41] | 15.4 [12.57 to 18.18] | 2.8 [1.00 to 4.63] | 6.2 [4.48 to 7.86]
  16 hrs Post-dose: number analyzed (Participants) | 32 | 33 | 32 | 35
  16 hrs Post-dose | 6.0 [2.65 to 9.35] | 8.9 [6.24 to 11.50] | -3.0 [-4.78 to -1.13] | 1.1 [-0.41 to 2.57]
  24 hrs Post-dose: number analyzed (Participants) | 32 | 34 | 33 | 33
  24 hrs Post-dose | 4.2 [2.28 to 6.14] | 6.2 [4.30 to 8.06] | -0.2 [-2.37 to 1.88] | 0.5 [-0.55 to 1.51]

ADVERSE EVENTS:
Time Frame: AE are collected during the entire study for each subject. From the Informed Consent Form (ICF) signature until end of study for each participant. The duration of each participant in the study was approximately 1 month. AE were followed until resolution or stabilization in case the event was ongoing at the end of study.
Arm/Group | All Subjects | 1.25 mg/kg Motixafortide | 2 mg/kg Motixafortide | Placebo SC | 400 mg Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36 | 0/37 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36 | 0/37 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 38/38 | 36/36 | 37/37 | 22/36 | 12/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=38) | 1.25 mg/kg Motixafortide (N=36) | 2 mg/kg Motixafortide (N=37) | Placebo SC (N=36) | 400 mg Moxifloxacin (N=36)
Leukocytosis (Blood and lymphatic system disorders) | 38 (72) | 36 (36) | 36 (36) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 5 (5) | 6 (6) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 13 (19) | 8 (8) | 10 (10) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 23 (30) | 9 (11) | 17 (17) | 0 (0) | 1 (2)
Injection site erythema (General disorders) | 37 (69) | 29 (33) | 28 (32) | 4 (4) | 0 (0)
Injection site hypoaesthesia (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 26 (34) | 15 (16) | 12 (13) | 5 (5) | 0 (0)
Injection site mass (General disorders) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 37 (159) | 32 (66) | 36 (82) | 10 (11) | 0 (0)
Injection site pruritus (General disorders) | 24 (42) | 17 (20) | 17 (19) | 3 (3) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 5 (7) | 0 (0) | 4 (6) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 16 (19) | 9 (9) | 7 (8) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 16 (23) | 11 (13) | 9 (10) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 15 (19) | 7 (7) | 11 (11) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5) | 4 (4) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Piloerection (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (53) | 21 (26) | 24 (26) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 26 (37) | 14 (14) | 22 (23) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 25 (32) | 10 (11) | 21 (21) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Injection site bruising (General disorders) | 7 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 14 (14) | 8 (8) | 4 (4) | 2 (2) | 0 (0)
Injection site haemorrhage (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 6 (6) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 11 (15) | 6 (6) | 4 (5) | 3 (3) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 4 (7) | 2 (3) | 4 (4) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 4 (6) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 8 (12) | 3 (3) | 6 (8) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (7) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 6 (10) | 4 (5) | 4 (5) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 2 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site necrosis (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT05293171/Prot_SAP_000.pdf